CLINICAL TRIAL: NCT01403792
Title: A Double-Blind, Placebo-Controlled, Randomised, Dose-Escalation Phase I Safety Study Of A Single Vaginal Administration Of P2G12 Antibody In Healthy Female Subjects
Brief Title: A Safety Study Of A Single Vaginal Administration Of P2G12 Antibody In Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRC282
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; Neutralising monoclonal antibody
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Up to 7mg P2G12 (Experimental)
  Interventions: Drug: P2G12
- Up to 14mg P2G12 (Experimental)
  Interventions: Drug: P2G12
- Up to 28mg P2G12 (Experimental)
  Interventions: Drug: P2G12
- Placebo (saline solution) (Placebo Comparator)
  Interventions: Drug: P2G12

INTERVENTIONS:
Drug: P2G12 — A single intravaginal administration of 1ml P2G12/placebo.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of intravaginal administration of P2G12. 11 subjects will receive P2G12/placebo. Three subjects in Group 1 will receive up to 7mg of P2G12, or placebo. Three subjects in Group 2 will receive up to 14mg of P2G12, or placebo and five subjects in Group 3 will receive up to 28mg of P2G12, or placebo. A safety review will take place before subjects in Groups 2 and 3 receive study drug to determine if it is safe to proceed to the next dose of P2G12. Vaginal and cervical inspections will be performed to determine what effect, if any, the study drug has had on the site of administration. Adverse event data will be collected throughout the trial.

DETAILED DESCRIPTION:
This is a phase I study in healthy women aged 18 to 50 years, which involves vaginal application of study drug P2G12 or placebo.

P2G12 is a monoclonal antibody (MAb) (a kind of protein), and belongs to a group of MAbs that can help to prevent and protect from HIV infection. Most of these MAbs have been produced using a system called Chinese Hamster Ovary cell (CHO-Cell) fermentation, e.g. C2G12. This method of production is very expensive and cannot produce enough MAbs on a scale required for the global market.

Unlike C2G12, P2G12 is manufactured from plants. It is hoped that plant manufacture of such MAbs may offer some solutions to the high cost and low output of CHO-cell fermentation.

This study is designed to confirm the safety of a vaginally delivered MAb (P2G12) derived from plants and manufactured to Good Manufacturing Practice (a quality standard used for the manufacture of medicinal products).

11 subjects will be enrolled consecutively in cohorts (groups); in each successive cohort a higher dose of study drug will be administered, as well as placebo. The dose range is from up to 7 to up to 28mg of P2G12 in saline.

Subjects attend 7 visits over 13 weeks. At visit 3 subjects receive a single administration of study drug/placebo. Study visits include the following procedures: physical exam, vital signs, blood and urine samples, cervical smear test and colposcopy (medical examination of the cervix).

The relationship of adverse events (AEs) and serious adverse events (SAEs) to P2G12 administration, and abnormal laboratory test results as compared to baseline (pre-dose) values, will determine the safety of P2G12 in the study.

Levels of P2G12 in vaginal and serum samples will be measured at particular time-points in order to understand how quickly P2G12 is broken down by the body (pharmacokinetics) and whether any P2G12 is absorbed into the systemic circulation.

ELIGIBILITY:
Inclusion Criteria:

* A female adult subject aged between 18 and 50 years old.
* They are in good health as determined by medical history, physical examination and clinical judgement before entering into the study.
* Subjects must agree to abstain from vaginal sexual intercourse for 72 hours before and after dosing.
* Subject must agree not to undertake any vaginal practices during study participation other than receptive intercourse with a male, or use of sanitary tampons during menses. Use of condoms without spermicidal agents is encouraged.
* Confirmation from the subject's GP that there is nothing in the subject's medical history that would prevent the subject from participating in the study.

Exclusion Criteria:

* They have a known or suspected ongoing vaginal disease, malignancy or abnormality (including non-menstrual vaginal discharge) discovered at time of screening.
* They have an abnormality, or non-menstrual discharge noted at screening colposcopy.
* They present in the samples obtained at the screening visit:

  1. positive results for HIV 1 or 2 antibody.
  2. positive results for Hepatitis B sAg, anti-Hepatitis C antibody
  3. positive syphilis serology
  4. positive test for Neisseria gonorrhoea or Chlamydia trachomatis on urine or urethral swab sample
  5. abnormal cervical smear cytology
* A clinically significant amount of protein or haemoglobin in the urine sample, determined by urine dipstick.
* They have received any form of immunosuppressive or immunomodulatory (e.g. vaccines) therapy in the past 6 months.
* They are receiving any medications via vaginal route.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Occurrence, intensity and relationship to P2G12 administration of local and general adverse events (AEs) throughout the study period after drug administration. | 35 days.

SECONDARY OUTCOMES:
Changes in levels of P2G12 in blood and vaginal secretions as compared to baseline. | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: Hubert A Bland, MBChB, Principal Investigator — University of Surrey
Locations (1):
- Surrey Clinical Research Centre, Guildford, Surrey, United Kingdom